CLINICAL TRIAL: NCT02027792
Title: Randomised Controlled Trial on the Efficacy of Cabbage Leaf Wraps in Symptomatic Primary Osteoarthritis of the Knee
Brief Title: Cabbage Leaf Wraps in Osteoarthritis of the Knee
Acronym: KoGon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Romy Lauche, Principle investigator, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-5581 KoGon
Record Dates: First submitted 2014-01-03; First posted 2014-01-06 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cabbage leaf wraps (Experimental): Daily application of cabbage leaf wraps over night, 4 weeks application
  Interventions: Other: Cabbage leave wraps
- Diclofenac gel (Active Comparator): daily application of diclofenac gel 4 weeks application
  Interventions: Drug: Diclofenac Gel
- Usual care (No Intervention): no specific intervention

INTERVENTIONS:
Other: Cabbage leave wraps
  Arms: Cabbage leaf wraps
Drug: Diclofenac Gel
  Arms: Diclofenac gel

SUMMARY:
This randomised controlled trial aims to investigate the efficacy of cabbage leaf cataplasms in the treatment of primary symptomatic osteoarthritis of the knee. 81 patients will be randomised into one of 3 groups and apply either cabbage leaf cataplasm or diclofenac gel daily for 4 weeks or receive only usual care. Efficacy will be measured using questionnaire on pain, disability, quality of life and pressure pain sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* osteoarthritis of the knee, Kellgren Lawrence stadium 2-3
* at least 50% of days with complaints
* initial pain intensity 45mm on a 100mm visual analoge scale

Exclusion Criteria:

* medication with corticoids or immunsupressing drugs
* secondary arthritis/arthrosis
* operation to the knee within 12 months prior
* injection within 4 weeks (cortison) or 6 months prior (hyaluronic acid)
* severe comorbidities (liver, kidney, asthma, psychiatric disorders etc.)
* participation in other studies
* pregnancy, breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 4 weeks
  pain intensity measured on three 0-100mm visual analog scales (actual, mean, worst pain)

SECONDARY OUTCOMES:
knee function (WOMAC) | 4 weeks
  physical everyday function using the validated WOMAC questionnaire
Quality of Life (SF-36) | 4 weeks
  health related quality of life with the validated SF-36 questionnaire
self-efficacy (ASES-D) | 4 weeks
  self-efficacy with the arthritis specific self efficacy scale in German
physical function (30second chair test) | 4 weeks
  validated test to measure how often patients can stand up from a chair in 30 seconds)
Pressure pain sensitivity | 4 weeks
  measured by an algometer at predefined areas
Adverse events | 4 weeks
  Safety measure
knee function (WOMAC) | 12 weeks
  physical everyday function using the validated WOMAC questionnaire
Quality of Life (SF-36) | 12 weeks
  health related quality of life with the validated SF-36 questionnaire
self-efficacy (ASES-D) | 12 weeks
  self-efficacy with the arthritis specific self efficacy scale in German
physical function (30second chair test) | 12 weeks
  validated test to measure how often patients can stand up from a chair in 30 seconds)
Pressure pain sensitivity | 12 weeks
  measured by an algometer at predefined areas
Adverse events | 12 weeks
  Safety measure
Pain intensity | 12 weeks
  pain intensity measured on three 0-100mm visual analog scales (actual, mean, worst pain)

OTHER OUTCOMES:
Course of Pain | 12 weeks
  measured by a diary including pain intensity on a visual analogue scale, medication
Satisfaction | 20 weeks
  Satisfaction with either treatments

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal and Integrative Medicine, Kliniken Essen-Mitte, Essen, Germany

REFERENCES:
- [Result] Lauche R, Graf N, Cramer H, Al-Abtah J, Dobos G, Saha FJ. Efficacy of Cabbage Leaf Wraps in the Treatment of Symptomatic Osteoarthritis of the Knee: A Randomized Controlled Trial. Clin J Pain. 2016 Nov;32(11):961-971. doi: 10.1097/AJP.0000000000000352. PMID 26889617